CLINICAL TRIAL: NCT02150161
Title: Fentanyl vs. Lidocaine/Ketamine Infusion for Hip Arthroscopy
Brief Title: Opioid vs. Opioid-free Anesthesia for Hip Arthroscopy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB estimated futility of the trial and safety risk
Sponsor: Clinica Santa Maria (Other)
Responsible Party: Principal Investigator, David Torres, Principal investigator, Clinica Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56csm2014001
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Opioid Free Anaesthesia; Postoperative Analgesia
MeSH Terms: interventions — Lidocaine; Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- lidocaine/ ketamine infusion (Experimental): lidocaine 1mg/Kg bolus, followed by continuous infusion 1 mg/kg/h AND ketamine 1mg/Kg bolus followed by continuous infusion 1 mg/kg/h
  Interventions: Drug: Lidocaine/ ketamine
- fentanyl (Active Comparator): iv fentanyl, 3ug/kg bolus
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Lidocaine/ ketamine
  Arms: lidocaine/ ketamine infusion
Drug: Fentanyl
  Arms: fentanyl

SUMMARY:
The purpose of this study is to determine whether an infusion of lidocaine/ketamine compared to fentanyl is equivalent in anesthesia effectiveness and can help reduce the incidence of postoperative nausea and vomiting in patients undergoing elective hip arthroscopy surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* ASA I-II
* Undergoing elective hip arthroscopy

Exclusion Criteria:

* Known allergies to study drugs
* Opioid use 1 month prior to surgery
* BMI >30
* Unable to comprehend visual analog scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting in the recovery room | first 3 postoperative hours
morphine consumption in the recovery room | first 3 postopeartive hours

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting on day 1 | 1st postoperative day
Anesthestic gas consumption | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: David Torres, MD; MSc, Principal Investigator — Clinica Santa Maria
Locations (1):
- Clinica Santa Maria, Santiago, Chile